CLINICAL TRIAL: NCT05810532
Title: Investigation on the Safety of 4-1 Hour Fasting Policy Before Sedation in Children.
Brief Title: NPO Before Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Eunah Cho, MD, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NPO1
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4H group (Active Comparator): fasting more than 4 hours before sedation
  Interventions: Other: 4 hours of fasting time
- 1H group (Experimental): oral hydration (water) is allowed 1 hour before sedation, while other food must be fasted more than 4 hours before sedation
  Interventions: Other: 1 hour of fasting time

INTERVENTIONS:
Other: 4 hours of fasting time — Oral intake is not allowed for 4 hours before sedation including water
  Arms: 4H group
Other: 1 hour of fasting time — Oral intake is not allowed for 4 hours before sedation, while water is allowed to intake before 1 hour of sedation
  Arms: 1H group

SUMMARY:
Pre-procedural fasting is routinely conducted to prevent pulmonary aspiration regarding sedation or anesthesia. However, prolonged fasting cause hypoglycemia, dehydration, nausea, and patient discomfort. Moreover, because children have small reserved energy, prolonged fasting need to be prohibited.

Therefore, this study is designed to investigate the safety and efficacy of new fasting policy allowing water until 1 hour before sedation compared to the standard fasting time (4 hours of fasting including water).

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for elective echocardiography
* Aged under 3 years old

Exclusion Criteria:

* Comorbidity other than hear disease or chromosomal disease
* Patients with delayed gastric emptying
* Patients with structural abnormalities of the stomach or esophagus
* Difficult airway management
* Parents refuse to participate in the study
* Unable to achieve sedation
* Neonatal

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Gastric astral cross-sectional area | 10 minutes before sedation
  Gastric astral cross-sectional area measured with gastric ultrasound

SECONDARY OUTCOMES:
Estimated gastric volume | 10 minutes before sedation
  Calculated gastric volume using the formula
Perlas grade | 10 minutes before sedation
  Perlas grade 0 : no risk of aspiration, Perlas grade 1 : minimal risk of aspiration, Perlas grade 2: high risk of aspiration
Quality of sdeation | 10 minutes after sedation
  0, no response to pain; 1, slight response to pain; 2, response to pain; 3, response to calling

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho E, Song J, Huh J, Kang IS, Kim HJ, Youn IY, Lee H, Kwak JH. Evaluation of Modified Fasting Protocols to Shorten Fasting Time Before Sedation in Children: A Prospective Randomized Noninferiority Trial. Paediatr Anaesth. 2025 Sep;35(9):753-760. doi: 10.1111/pan.15142. Epub 2025 Jun 18. PMID 40530767